CLINICAL TRIAL: NCT01660009
Title: Adverse Effects of Systemic Hypoglycemia Exposure on Endothelial Function in Humans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Funding
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MCW-MEW3
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2015-04

CONDITIONS: Type 2 Diabetes
Keywords: Endothelial Function; Hypoglycemia; Mitochondria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoglycemia First (Experimental): Individuals will undergo a hyperinsulinemic hypoglycemic clamp in their 1st study visit after passing screening, and a euglycemic clamp in their second visit.
  Interventions: Other: Glycemic clamping
- Euglycemia First (Experimental): Individuals will undergo a hyperinsulinemic euglycemic clamp in their 1st study visit after passing screening, and a euglycemic clamp in their second visit.
  Interventions: Other: Glycemic clamping

INTERVENTIONS:
Other: Glycemic clamping — During hypoglycemic clamping, individuals will have a blood glucose level of 50-60 mg/dL for approximately 1 hour prior to outcome measurements. During euglycemic clamping, individuals will have a blood glucose level of 85-99 mg/dL for approximately 1 hour prior to outcome measurements.

SUMMARY:
Prior work suggests exposure to low glucose levels (hypoglycemia) is associated with increased cardiovascular risk. However, whether there is a causal relationship between cardiovascular events and hypoglycemia remains unclear with conflicting data in the literature. In this study, we plan to study whether acute exposure of patients to clinically relevant (50-60 milligrams/deciliter) levels of hypoglycemia induces or worsens blood vessel endothelial dysfunction- a key 1st step in the development of heart attacks and strokes. This will be determined in humans both with and with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

- Type 2 Diabetes Inclusion Criteria

1. Adult age 21 or older
2. If on 3-hydroxy-3-methyl-glutaryl-coenzyme A reductase reductase therapy, must be on a stable dose for at least 6 weeks prior to enrollment
3. Diagnosis of type 2 diabetes by a physician as defined by the American Diabetes Association standard criteria: 1) Fasting Plasma glucose at or above 126 mg/dL 2) a two-hour value in an oral glucose tolerance test at or above 200 mg/dL, or 3) a random plasma glucose concentration 200 mg/dL in the presence of symptoms, or 4) glycosylated hemoglobin greater than or equal to 6.5%.

Score of < 4 using the Gold method for assessing hypoglycemia awareness

Inclusion Criteria for Healthy subjects

1. Adult age 21 or older
2. No evidence of metabolic syndrome or diabetes, hypertension (BP≥140/90), or high cholesterol (LDL≥160) at the time of screen.

Exclusion Criteria:

1. History of stroke, peripheral arterial disease, or coronary artery disease (as defined by the presence of at least one coronary stenosis ≥ 40% on angiography or by confirmed history of myocardial infarction by standard criteria)
2. Evidence of other evident major illness including chronic renal insufficiency(plasma creatinine > 1.4 for women or 1.5 for men), liver disease (aspartate aminotransferase or alanine aminotransferase greater than 2.5 x normal), and cancer currently undergoing therapy or had therapy for cancer within 1 year of enrollment.
3. Pregnancy as determine by urinary pregnancy test
4. Subjects on warfarin, oral anti-thrombin inhibitors, or thienopyridines
5. Subjects who have had changes to dosing of thiazolidinedione, dipeptidyl peptidase-4 (DPP-4) inhibitor, or metformin therapy within 6 weeks of enrollment.
6. Failed Allen's test in both arms - unable to safely place an arterial line
7. Glucose reading of < 50 mg/dL and/or episodes of symptomatic hypoglycemia requiring the assistance of another person for recovery in the 2 years prior to enrollment.
8. History of hypoglycemic convulsions
9. Current fluoxetine therapy (known to interfere with neuroendocrine response to hypoglycemia)
10. Glycosylated hemoglobin over 8.5%
11. On aldosterone antagonist therapy at the time of enrollment
12. On insulin therapy at the time of screening.
13. History of allergy to local anesthetic injection like lidocaine.
14. Age below 21.

Exclusion Criteria for Healthy Subjects:

1. Meet any of the exclusion criteria for diabetic or metabolic syndrome group Meet criteria for type 2 diabetes or metabolic syndrome
2. On medication for cholesterol or blood pressure.
3. History of allergy to local anesthetic injection like lidocaine.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Flow induced Dilation of the Brachial Artery (FMD%) | 1 hour

SECONDARY OUTCOMES:
Measurement of total and phosphorylated endothelium-derived NO synthase expression in radial artery endothelial cells. | 1 hour
Measurement of mitochondrial membrane potential | 1 hour
  Performed on captured radial artery endothelial cells.
Mitochondrial superoxide production | 1 hour
  From capture radial artery endothelial cells.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Widlansky, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States